CLINICAL TRIAL: NCT06306742
Title: Open-label Placebo in Manual Therapies: a Pilot Study.
Brief Title: Open-label Placebo in Manual Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Studio Osteopatico Busto Arsizio (Other)
Responsible Party: Principal Investigator, Carolina Lavazza, Principal investigator, Studio Osteopatico Busto Arsizio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ct9874
Record Dates: First submitted 2024-02-29; First posted 2024-03-12 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2024-03

CONDITIONS: Low Back Pain, Recurrent
Keywords: Placebo; Placebo effect; Open-label trial
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- OMT (Active Comparator): Participants will receive manual treatments. The treatment will include soft-tissue, joint mobilization techniques of the lumbar and sacral region. The treatment will also include the approach of the abdomen and lower limb with the same type of techniques.
  Four treatments will be provided at 1, 2, 4 and 8 weeks.
  Interventions: Other: Osteopathic manipulative treatment
- Open-label placebo (Experimental): This group will receive an open-label placebo. The manual treatment will be performed in the same areas of the active comparator but using a very light pressure. Additionally, before the start of the treatment, Four treatments will be provided at 1, 2, 4 and 8 weeks.
  Interventions: Other: Open-label placebo
- Waiting list (No Intervention): Participants will receive no treatment.

INTERVENTIONS:
Other: Open-label placebo — Light pressure manual therapy
  Arms: Open-label placebo
Other: Osteopathic manipulative treatment — Manual therapy
  Arms: OMT

SUMMARY:
to investigate the effects of placebo in patients affected by low-back pain.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (+18 years) who complain of chronic non-specific low back pain for at least 3 months with or without pain exacerbations at the time of recruitment, will be included.

-Patients will need to have a diagnosis of low back pain made by a physician

Exclusion Criteria:

* pathologies such as ankylosing spondylitis, infections, fractures, tumors or metastases.
* Pregnant women
* patients with previous spinal surgery or undergoing cortisone therapy in the 6 months prior to the trial
* diseases that may affect the interpretation of results such as fibromyalgia
* patients currently being treated by other specialists or other manual therapists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Change in Numeric Rating Scale | Change from baseline of numeric rating scale at week 2, 4 and 8.
  a verbal determination of a pain level on a scale from 0 to 10, in which 0 represents no pain and 10 represents excruciating pain.
Adverse effects | through study completion (8 weeks)
  Number and types of adverse effects occurred after intervention

SECONDARY OUTCOMES:
Change in measures of Von Frey filaments | from baseline at week 2,4 and 8.
  Changes in pressure measures
Changes in algometer measurements | from baseline at week 2, 4 and 8
  Changes in pressure with algometer
Use of analgesics | The week before the scheduled visit.
  Usage (Yes/no), number and type of analgesics used

CONTACTS AND LOCATIONS:
Locations (1):
- CTFO, Saronno, Varese, Italy

IPD SHARING:
Plan to Share IPD: No